CLINICAL TRIAL: NCT05711498
Title: Non-invasive Investigation of Excitability Changes in the Human Spinal Cord: the Effect of Transcutaneous Spinal Direct Current Stimulation (tsDCS) on Nociceptive Flexion Reflexes
Brief Title: Non-invasive Modulation of Spinal Cord Nociceptive Reflexes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Max Planck Research Group Pain Perception (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PP016
Record Dates: First submitted 2022-12-10; First posted 2023-02-03 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anodal thoracic tsDCS (Experimental): Anodal tsDCS will be applied over the T12 vertebra
  Interventions: Other: Transcutaneous spinal direct current stimulation (tsDCS)
- Cathodal thoracic tsDCS (Experimental): Cathodal tsDCS will be applied over the T12 vertebra
  Interventions: Other: Transcutaneous spinal direct current stimulation (tsDCS)
- Sham thoracic tsDCS (Sham Comparator): Sham tsDCS will be applied over the T12 vertebra
  Interventions: Other: Transcutaneous spinal direct current stimulation (tsDCS)

INTERVENTIONS:
Other: Transcutaneous spinal direct current stimulation (tsDCS) — tsDCS will be carried out using a direct current stimulator (DC-Stimulator Plus, neuroConn, Ilmenau, Germany), with one electrode placed above the thoracic spinal cord and the other electrode placed on the right shoulder. We will employ rectangular electrodes of 7 x 5 cm size (neuroConn, Ilmenau, Germany) covered by electrode paste (Ten20 Conductive Paste, Weaver and Company, Aurora, USA). Stimulation will consist of the following phases: a fade-in period of 15 seconds, a plateau period of 20 minutes (with stimulation at 2.5mA either anodally or cathodally) and a fade-out period of 15 seconds. Sham stimulation will follow the anodal montage with 15-second fade-in and fade-out periods, but only 45 seconds of plateau stimulation at 2.5 mA. Such a combination of stimulation and electrodes results in a current density of 0.071mA/cm2, well below thermal and histological limits for current density.

SUMMARY:
The aims of this study are threefold. First, to investigate whether spinal nociceptive processing - represented here by the nociceptive flexion reflex (NFR) - is influenced by thoracic transcutaneous spinal direct current stimulation (tsDCS) in a spatially selective manner, i.e., whether effects are only observed for lower limb NFRs, but not for upper limb NFRs. Second, to investigate - in a double-blind, sham-controlled, within-participant design - whether anodal and cathodal tsDCS do affect the NFR in a polarity-dependent manner. Third, to investigate whether tsDCS effects observed on a spinal measure (NFR) are also observed in responses that are mediated supra-spinally, namely autonomic parameters and pain intensity ratings.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers between the ages of 18 and 40 years
2. Having participated in the MRI medical assessment session and consented to taking part in 3T MRI measurements in written form
3. Having participated in the magnetic/electric neurostimulation medical assessment session and consented to taking part in magnetic/electric neurostimulation experiments in written form
4. Voluntary participation and signing of the study-specific consent form

Exclusion Criteria:

1. Existence of any contraindications for MRI measurements and magnetic/electric neurostimulation experiments
2. Pregnancy or breastfeeding
3. Very dry or sensitive skin (e.g., intolerance to creams/shampoos)
4. Chronic skin diseases - such as eczema or neurodermatitis - in the area of somatosensory / nociceptive stimulation (arm or hand, leg or foot) or electrophysiological data recording (upper body, arm, leg)
5. Scar tissue in the area of somatosensory / nociceptive stimulation (arm or hand, leg or foot) or electrophysiological data recording (upper body, arm, leg)
6. Acute sunburn in the area of somatosensory / nociceptive stimulation (arm or hand, leg or foot) or electrophysiological data recording (upper body, arm, leg)
7. Current or recurring pain
8. Injuries to the nervous system
9. History of or current neurological or psychiatric disorders
10. Chronic diseases that require permanent medication (e.g., asthma, diabetes mellitus, etc.)
11. Persons not capable of giving consent (e.g., in case of dementia)
12. Lack of consent with regards to report of incidental findings

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in NFR amplitude | Baseline and immediately after the intervention
  90-150ms for lower limb, 60-200ms for upper limb
Change in pain intensity rating | Baseline and immediately after the intervention
  One rating per trial on a standard visual analogue scale (VAS); internally numbered from 0 (no sensation) to 100 (unbearable pain)
Change in skin conductance response | Baseline and immediately after the intervention
  Amplitude maximum before onset of pain rating
Change in heart period acceleration | Baseline and immediately after the intervention
  Amplitude maximum before onset of pain rating

SECONDARY OUTCOMES:
Change in NFR area | Baseline and immediately after the intervention
  90-150ms for lower limb, 60-200ms for upper limb

CONTACTS AND LOCATIONS:
Locations (1):
- Max Planck Research Group Pain Perception, Leipzig, Germany

IPD SHARING:
Plan to Share IPD: No